CLINICAL TRIAL: NCT06083948
Title: Vasopressor Impact on Brain Circulation, Organ Blood Flow and Tissue Oxygenation During Anesthesia in Neurosurgical Patients
Brief Title: Vasopressor Impact on Brain Circulation, Organ Blood Flow and Tissue Oxygenation During Anesthesia
Acronym: IMPACT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMPACT study
Record Dates: First submitted 2023-09-26; First posted 2023-10-16 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noradrenaline (Experimental): Noradrenaline
  Interventions: Drug: Noradrenalin
- Phenylephrine (Active Comparator): Phenylephrine
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Noradrenalin — Infusion of noradrenaline during anesthesia and surgery
  Other Names: Noradrenaline
  Arms: Noradrenaline
Drug: Phenylephrine — Infusion of phenylephrine during anesthesia and surgery
  Other Names: metaoxedrin
  Arms: Phenylephrine

SUMMARY:
The optimal vasopressor for ensuring organ blood flow and tissue oxygen delivery during surgery remains undetermined. This study aim to compare the effects of noradrenaline vs. phenylephrine infusion on blood flow and oxygen delivery to the brain and various other organs in anesthetized neurosurgical patients.

DETAILED DESCRIPTION:
The brain and other blood flow sensitive organs are vulnerable to hypotension during neurosurgery. As a countermeasure, vasopressor agents are often administered to increase blood pressure. The ultimate goal of the vasopressor is to secure perfusion of vital organs and fulfill their metabolic demand. However, the optimal vasopressor for ensuring organ blood flow and tissue oxygen delivery during surgery remains undetermined.The aim of this study is to compare the effects of noradrenaline vs. phenylephrine infusion on blood flow and oxygen consumption in the brain and various other organs in anesthetized neurosurgical patients.

The project constitutes a clinical randomized study involving 32* patients diagnosed with brain tumors. The study is conducted on the same day as their scheduled brain tumor surgery. The study is designed as a randomized, double-blinded clinical trial, with two distinct groups: Group 1 receives phenylephrine, while Group 2 receives noradrenaline.

PET exams of blood flow and oxygen consumption in brain and organs(including myocardium, kidney, liver, spinal cord, organs supplied by the splanchnic circulation, muscle tissue and other organs) are performed using a PET scanner with a wide field of view. The wide field of view allow for simultaneous multiorgan blood flow and oxygen consumption measurements.

Four positron emission tomography (PET) examinations are performed prior to the surgical procedure. The first PET examination (PET 1) is performed on the awake patient. The patient is then anesthetized, and the PET exam is repeated (PET 2). Vasopressor infusion is initiated and titrated to increase mean arterial blood pressure(MABP) above 60 mmHg, or by 10% relative to baseline(baseline MABP is measured prior to PET 2). The PET exam is repeated (PET 3). MABP is further increased to above 70 mmHg or by 20 % relative to the baseline level and the PET exam is repeated (PET 4). The anesthetized patient is then transported to the surgical theatre and surgery is initiated. During the surgical procedure, MABP is maintained between 70-80 mmHg according to institutional guidelines. The vasopressor infusion is terminated after completion of the surgery.. Invasive blood pressure, cardiac output (CO),depth of anesthesia (bispectral index) and brain tissue oxygen saturation(near infrared spectroscopy) are continuously measured.An MRI examination is performed 24 hours after surgery to detect any ischemic lesions possibly associated with the vasopressor infusion.

* The initial sample size of 40 patients was reduced to 32 patients in april 2024 (after inclusion of 4 patients). The change in sample size is due to unexpected limited scanner availability and unexpected difficuties with patient recruitment. These factors will be associated with a longer period of patient inclusion and consequently longer time before study completion which we find unacceptable.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of supratentorial malignant or non-malignant brain tumors. Preferably 3 cm or larger( measured as the largest diameter in any plane on MRI).
2. Scheduled for elective supratentorial craniotomy.
3. Patients aged between 18 and 75 years.
4. American Society of Anesthesiologists status 1-3

Exclusion Criteria:

1. History of allergy or intolerance to one of the study medications.
2. Active treatment with monoamine oxidase inhibitors.
3. An American Society of Anesthesiologists (ASA)physical status IV-VI.
4. Pregnancy or breastfeeding.
5. Inability to provide written informed consent -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | Up to 3 hours (measured on the day of surgery prior to the surgical procedure)
  Blood flow measured in milliliters per minute through selected regions of the brain as determined by Positron Emission Tomography

SECONDARY OUTCOMES:
Cerebral metabolic rate of oxygen | Up to 4 hours (measured on the day of surgery prior to the surgical procedure)
  Cerebral oxygen consumption in selected regions of the brain as determined by Positron Emission Tomography
Blood flow through body organs in milliliters per minute as determined by Positron Emission Tomography | Up to 4 hours (measured on the day of surgery prior to the surgical procedure)
  Blood flow in various body organs supplied by the systemic circulation
Blood pumped out by the heart per minute (cardiac output) | Up to one day
  Cardiac output as determined by Positron Emission Tomography and/or by beat-to-beat determination by analysis of the arterial blood pressure waveform
Ischemic lesions | Up to 3 days
  Ischemic lesions possibly associated with vasopressor use as detected on the postoperative MRI examination
Cerebral tissue oxygen saturation | Up to one day
  Cerebral tissue oxygen saturation as measured with near infrared spectroscopy (NIRS)
Bispectral Index (BIS) | Up to one day
  Depth of anesthesia as measured by BIS
Organ metabolic rate of Oxygen | Up to 3 hours (measured on the day of surgery prior to the surgical procedure)
  Oxygen consumption in various organs as measured by Positron Emission Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Mads Rasmussen, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
THe trial data may be shared upon request to the Investigator
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Other researchers may request the data after publication of the primary results and for a period of 10 years
Access Criteria: No specific criteria

REFERENCES:
- [Derived] Faisal Mohamad N, Koch KU, Aanerud J, Meier K, Mikkelsen IK, Espelund US, Eriksen CF, Juul N, Alstrup KB, Jespersen B, Fries LM, Tankisi A, Dyrskog S, Cortnum SOS, Sindby AK, Borghammer P, Tolbod LP, Meng L, Korshoej AR, Rasmussen M. Impact of norepinephrine versus phenylephrine on brain circulation, organ blood flow and tissue oxygenation in anaesthetised patients with brain tumours: study protocol for a randomised controlled trial. BMJ Open. 2025 Mar 25;15(3):e095172. doi: 10.1136/bmjopen-2024-095172. PMID 40132839